CLINICAL TRIAL: NCT03212053
Title: Prospective Study of Different Biological Tests (Multiplate, ROTEM) in a Cohort of Patients Followed for Essential Thrombocytemia (ET)
Acronym: THETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 69HCL17_0091; 2017-A00737-46 (Other: ANSM)
Record Dates: First submitted 2017-06-30; First posted 2017-07-11 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Thrombocythemia Essential
Keywords: Essential thrombocythemia; Multiplate; ROTEM; haemorrhage; thrombosis; Vasodilatator Stimulated Phosphoprotein (VASP)
MeSH Terms: conditions — Thrombocythemia, Essential; Hemorrhage; Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Essential Thrombocythemia (Other): patients who come in consultation at diagnosis or during the follow-up for an Essential Thrombocythemia.
  They will have biological tests of haemostasis at each consultation (Multiplate, ROTEM, VASP)
  Interventions: Biological: biological tests of haemostasis at each consultation (Multiplate, ROTEM, VASP)

INTERVENTIONS:
Biological: biological tests of haemostasis at each consultation (Multiplate, ROTEM, VASP) — Patients will have blood samples at each consultation (2 or 3 sampling tubes) in order to carry out systematically three biological tests

SUMMARY:
There is no prospective study published on the Essential Thrombocythemia and the correlation between this specific disease, its complications and the biological variations observed.

The aim of this study is to demonstrate a correlation between biological tests of haemostasis, as Multiplate analyser and thromboelastometry (ROTEM) and the occurrence of clinical complications, thrombosis and/or haemorrhage, in order to determine if this biological tests could be biological prognostic factors

ELIGIBILITY:
Inclusion Criteria:

* Adult aged more than 18 years old
* Patient followed in consultation for an Essential Thrombocythemia at diagnosis or during the follow-up
* Collection of the informed consent
* Patient affiliated to Social Security

Exclusion Criteria:

* Patients aged less than 18 years old
* Refusal of signature of the informed consent
* Patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of thrombotic complications | every 4 months, up to 18 months
  All thrombotic complications will be gathered by the investigators during the four months following the realization of Multiplate and ROTEM test
Occurrence of haemorrhagic complications | every 4 months, up to 18 months
  All haemorrhagic complications will be gathered by the investigators during the four months following the realization of Multiplate and ROTEM test

SECONDARY OUTCOMES:
Occurrence of thrombotic complications | every 4 months, up to 18 months
  All thrombotic complications will be gathered by the investigators during the four months following the realization of VASP test
Occurrence of haemorrhagic complications | every 4 months, up to 18 months
  All haemorrhagic complications will be gathered by the investigators during the four months following the realization of VASP test
Changes of tests results according to medical treatments | every 4 months, up to 18 months
  All modifications of medical treatments will be gathered at each consultation to analyse changes of biological tests results
Description of platelet physiopathology | the day of inclusion
  Using a specific test of release of ATP to study the platelet physiopathology in Essential Thrombocythemia only for patients seen at diagnosis and naive of all medical treatment
Description of platelet physiopathology | the day of inclusion
  Using electronic microscopy to study the platelet physiopathology in Essential Thrombocythemia only for patients seen at diagnosis and naive of all medical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fiorenza BARRACO, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France